CLINICAL TRIAL: NCT03086954
Title: Open, Single Arm,Multicenter Phase 2 Clinical Study to Evaluating the Efficacy and Safety of the Chimeric Antigen Receptor T Cell Immunotherapy (CAR-T) for CD19 Positive Lymphoma
Brief Title: Study Evaluating the Efficacy and Safety With CAR-T Immunotherapy for CD19 Positive Lymphoma
Acronym: EECPL
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sinobioway Cell Therapy Co., Ltd. (Industry)
Collaborators: Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WM-CART-02
Record Dates: First submitted 2017-03-13; First posted 2017-03-22 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Lymphoma
Keywords: CD19 positive lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): Name:The Chimeric Antigen Receptor T Cell Immunotherapy (CAR-T) Dosage form：injection Dosage:100ml/time Frequency:The first day,the second day,29 days,injection once a day in this three days Duration:Only injection three times
  Interventions: Biological: The Chimeric Antigen Receptor T Cell Immunotherapy (CAR-T)

INTERVENTIONS:
Biological: The Chimeric Antigen Receptor T Cell Immunotherapy (CAR-T) — This study have only one arm that is CAR-T experimental arm. Firstly all participators will be attended the screening, who passed the screening for the treatment of CAR-T cells, the CAR-CD19-modified T cells can recognize and kill tumor cells in the body，follow-up 35 months.

SUMMARY:
This open, single-arm,multicenter 2 phase clinical study will treat the patient who have CD19 positive lymphoma with an infusion of the patient's own T cells that have been genetically modified to express a chimeric antigen receptor(CAR)that will bind to tumour cells modified to express the CD19 protein on the cell surface. The study will determine if these modified T cells help the body's immune system eliminate tumour cells .The trial will also study the safety of treatment for CAR-T, how long CAR-T cells stay in the patient's body and the impact on this treatment for survival.

DETAILED DESCRIPTION:
This is an open, single-arm,multicenter 2 phase clinical study to evaluate efficacy and safety of chimeric antigen receptor T cell immunotherapy (CAR-T) in the treatment of CD19 positive lymphoma. The study will be conducted using a phaseⅠ/Ⅱdesign the study will have the following sequential phases: part A (screening, leukapheresis, cell product preparation and cytoreductive chemotherapy) and part B (treatment and follow-up). The follow-up period for each participant is approximately 35 months after the final CAR-T infusion. The total duration of the study are expected to be approximately 3 years. A total of 24 patients may be enrolled over a period of 3 years.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age older than 16 years old,gender and race no limited.
* 2.Pathological diagnosis of CD19 express positive recurrent or refractory B lymphoma, satisfy any of the following a diagnosis of recurrent or refractory lymphoma: (1) According to the standard solution standardization more than four courses of treatment, tumor size < 50% or progression;(2) According to the standard solution treatment of complete remission, after recurrence again with the original plan or the national expert consensus recommended second-line cannot again get to complete remission (3) Relapse after hematopoietic stem cell transplantation.
* 3.Patients into the group needs lesions to be available for testing or evaluating disease.
* 4.ECOG score reaches 0 to 1 points.
* 5.Patients into the group of White Blood Cell counts in peripheral blood acuity≥ 1.0 x10^9 / L.
* 6.Estimated survival times > 90 days.
* 7.Patients have self-knowledge ability, can sign the informed consent form.

Exclusion Criteria:

* 1.Pregnant or lactating women.
* 2.Uncontrolled infection.
* 3.HIV infection, hepatitis B or C activity period.
* 4.Patients who need long-term immunosuppressive therapy (Such as allergies, autoimmune diseases, GVHD, etc.)
* 5.Combined activity of the central nervous system malignant tumor invasion.
* 6.Abnormal coagulation function, patients with severe thrombosis.
* 7. Organ failure Heart：class Ⅱ or above. Liver：class Ⅱ or above( Refer to Classification of Wuhan Conference (1983)). Kidney: The second stage of renal insufficiency or above. Lung: class Ⅱdecreased slightly or above. Brain: The central nervous system transfer or have active lesions.
* 8.Patients who have participated in other clinical trials in the past 30 days or or participate in other clinical trials at the same time.
* 9.Investigator believe that the patient is not suitable to participate in the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-04 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
The objective reaction rate of patients with CD19 positive lymphoma after autologous CAR-T cell therapy. | up to 90 days
  The objective reaction rate will be determined by the evaluation of CT/PET-CT.Evaluation of the objective reaction rate according to the non-hodgkin's lymphoma curative effect evaluation criteria of international lymphoma group. The objective reaction rate = (complete remission (CR) number + partial remission (PR) number / total number of cases receiving treatment.

SECONDARY OUTCOMES:
Progression free survival time | 3years
  From patients into the group to the interval between disease progression or death.
Overall survival time | 3years
  From all patients into the group to the interval between death caused by any reason .
Patients - -based Quality of Life Evaluation | 3years
  According to the EORTC quality of life of the core scale criteria QLQ-C30(V3.0) to evaluate patients life quality.
3°or above incidence rate of serious adverse reaction related to treatment | 3years
  According to CTCAE v4.0 to evaluate incidence rate of serious adverse reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Jifeng Feng, Professor, Principal Investigator — Director of medical oncology
Locations (1):
- Jiangsu Cancer hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Turtle CJ, Hanafi LA, Berger C, Hudecek M, Pender B, Robinson E, Hawkins R, Chaney C, Cherian S, Chen X, Soma L, Wood B, Li D, Heimfeld S, Riddell SR, Maloney DG. Immunotherapy of non-Hodgkin's lymphoma with a defined ratio of CD8+ and CD4+ CD19-specific chimeric antigen receptor-modified T cells. Sci Transl Med. 2016 Sep 7;8(355):355ra116. doi: 10.1126/scitranslmed.aaf8621. PMID 27605551
- See also: Immunotherapy of non-Hodgkin's lymphoma with a defined ratio of CD8+ and CD4+ CD19-specific chimeric antigen receptor-modified T cells. — https://www.ncbi.nlm.nih.gov/pubmed/27605551